CLINICAL TRIAL: NCT06624852
Title: Clinical Validation of PROPECG-TMT: Evaluation of Ability of the Artificial Intelligence Model, PROPECG-TMT, to Improve Physician's in Screening Patients Who Needs Coronary Artery Revascularization Based on TMT-ECG.
Brief Title: Clinical Validation of PROPECG-TMT
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2023-0086
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Performances with AI assistance: Performances of screening coronary artery revascularization with PROPECG-TMT
  Interventions: Other: Screening for coronary artery revascularization based on TMT-ECG
- Performances without AI assistance: Performances of screening coronary artery revascularization without PROPECG-TMT
  Interventions: Other: Screening for coronary artery revascularization based on TMT-ECG

INTERVENTIONS:
Other: Screening for coronary artery revascularization based on TMT-ECG — Screening for coronary artery revascularization based on TMT-ECG with and without the assistance of PROPECG-TMT

SUMMARY:
This clinical validation evaluates the performances of physicians with and without learning with PROPECG-TMT assistance for screening coronary artery revascularization on TMT-ECG.

There are two endpoints used to evaluate performances: Accuracy (primary endpoints with pair specificity/sensitivity, and PPV/NPV), and time needed for screening (secondary endpoints with time measurements in all cases).

ELIGIBILITY:
Inclusion Criteria:

* TMT ECG exams adjudicated as equivocal cases

Exclusion Criteria:

* Exams not converting to median beat ECG
* Exams not containing interpretable exercise

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * At least 100 TMT ECG exams adjudicated as equivocal cases
  * 7% of exams are positive (one or more percutaneous coronary interventions or coronary artery bypass surgeries have been performed) and 93% of exams are negative (no percutaneous coronary interventions or coronary artery bypass surgery have been performed)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
measurement of screening performances | 1 month
  calculation of sensitivity, specificity, NPV, PPV

SECONDARY OUTCOMES:
Time needed for screening all cases | 1 month
  measurement of the time and comparison between the two cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedicine Systems Informatics, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No